CLINICAL TRIAL: NCT05432635
Title: Pilot/Feasibility Study of CMV-Specific CD19-CAR T Cells Plus CMV-MVA Triplex Following Autologous Hematopoietic Stem Cell Transplantation for Patients With Intermediate or High Grade B-Lineage Non-Hodgkin Lymphoma (B-NHL)
Brief Title: Genetically Modified T-cells (CMV-Specific CD19-CAR T-cells) Plus a Vaccine (CMV-MVA Triplex) Following Stem Cell Transplantation for the Treatment of Intermediate or High Grade B-cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20695; NCI-2022-04622 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20695 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH); P50CA107399 (NIH)
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: B-Cell Non-Hodgkin Lymphoma; Diffuse Large B-Cell Lymphoma; Mantle Cell Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Transformed Non-Hodgkin Lymphoma; Transformed Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — Bone Marrow Purging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CMV-specific CD19-CAR T cells, triplex vaccine) (Experimental): CONDITIONING REGIMEN: Patients receive standard conditioning regimen (typically carmustine, etoposide, cytarabine, melphalan) beginning approximately on day -9 in the absence of disease progression or unacceptable toxicity.
  TRANSPLANTATION: Patients undergo autoHSCT on day -2.
  CAR T-CELLS AND VACCINATION: Patients receive CMV-specific CD19-CAR T cells IV on day 0 and CMV-MVA triplex vaccine IM on days 28 and 56 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-CD19-CAR CMV-specific T-lymphocytes; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine; Procedure: Myeloablative Conditioning

INTERVENTIONS:
Biological: Anti-CD19-CAR CMV-specific T-lymphocytes — Given IV
  Other Names: CMV-specific CD19-CAR T Cells (SY); CMV-specific CD19 CAR-T Cells (SY); Anti-CD19-CAR CMV-specific T-cells (SY)
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autoHSCT
Biological: Multi-peptide CMV-Modified Vaccinia Ankara Vaccine — Given IM
Procedure: Myeloablative Conditioning — Given standard conditioning regimen

SUMMARY:
This phase I trial studies the safety and side effects of cytomegalovirus (CMV) specific CD19-chimeric antigen receptor (CAR) T-cells along with the CMV-modified vaccinia Ankara (MVA) triplex vaccine following a stem cell transplant in treating patients with high grade B-cell non-Hodgkin lymphoma. CAR T-cells are a type of treatment in which a patient's T-cells (a type of immune system cell) are changed in the laboratory so they will attack cancer cells. T-cells are taken from a patient's blood. Then the gene for a special receptor that binds to a certain protein on the patient's cancer cells is added in the laboratory. The special receptor is called a chimeric antigen receptor (CAR). Large numbers of the CAR T-cells are grown in the laboratory and given to the patient by infusion. Vaccines such as CMV-MVA triplex are made from gene-modified viruses and may help the body build an effective immune response to kill cancer cells. Giving CMV-specific CD19-CAR T-cells plus the CMV-MVA triplex vaccine following a stem cell transplant may help prevent the cancer from coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the safety and describe the toxicity profile of anti-CD19-CAR CMV-specific T-lymphocytes (CMV-specific CD19-CAR T cells) alone and when given in combination with multi-peptide CMV-modified vaccinia Ankara vaccine (CMV-modified vaccinia Ankara [MVA] triplex vaccine) following autologous hematopoietic cell transplantation (autoHSCT) to treat participants with intermediate or high grade B-lineage non-Hodgkin lymphoma (NHL) who are in first relapse after achieving complete remission (CR) or did not achieve CR after a first line therapy.

SECONDARY OBJECTIVES:

I. Determine the feasibility of autologous CMV-specific CD19-CAR T cell manufacturing, as assessed by the ability to meet the required cell dose and product release requirements in 5 out of 6 enrolled participants.

II. Determine short- and longer-term CMV-specific CD19-CAR T cell in vivo expansion and persistence.

III. Assess whether the CMV-specific CD19-CAR T cells respond to CMV-MVA triplex vaccine.

IV. Estimate the rate of CMV reactivation after CAR T cell infusion. V. Estimate the rate of progression-free survival (PFS) and median overall survival (OS) at 12 months post-autoHSCT.

EXPLORATORY OBJECTIVES:

I. Assess whether the CMV-specific CD19-CAR T cells respond to CMV-MVA triplex vaccine when administered to participants that received CAR T cells only in the safety lead-in portion in the expansion phase of the study (i.e., once safety of the CMV-MVA triplex vaccine is established in the feasibility portion of the study).

Ia. Participants who receive CMV-specific CD19-CAR T cells in the safety lead-in portion of the study may be eligible to receive the CMV-MVA Triplex vaccine in the expansion portion of the study per principal investigator (PI) discretion and if all other criteria to proceed with vaccine administration are met.

OUTLINE:

CONDITIONING REGIMEN: Patients receive standard conditioning regimen (typically carmustine, etoposide, cytarabine, melphalan) beginning approximately on day -9 in the absence of disease progression or unacceptable toxicity.

TRANSPLANTATION: Patients undergo autoHSCT on day -2.

CAR T-CELLS AND VACCINATION: Patients receive CMV-specific CD19-CAR T cells intravenously (IV) on day 0 and CMV-MVA triplex vaccine intramuscularly (IM) on days 28 and 56 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 18-24 hours, weeks 1-3, at 1 month, at day 84, months 4-11, and at 1 year. Patients with disease progression or starting a prohibited therapy are also followed up on months 2-4, 6, and 12 after CAR T cell infusion, and then yearly for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative.

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies.

  * If unavailable, exceptions may be granted with study PI approval
* Note: For research participants who do not speak English, a short form consent may be used with a City of Hope (COH) certified interpreter/translator to proceed with screening and leukapheresis, while the request for a translated full consent is processed
* Age >= 18 years
* Karnofsky performance status (KPS) >= 70
* Life expectancy >= 16 weeks at the time of enrollment
* Patients with an indication to be considered for HSCT, who are diagnosed with intermediate or high-grade B cell NHL (e.g., diffuse large B-cell lymphoma [DLBCL], mantle cell lymphoma [MCL], or transformed NHL) in first relapse after achieving complete remission (CR) or did not achieve CR after a first line therapy

  * Note: COH pathology review should confirm that research participant's diagnostic material is consistent with history of intermediate or high-grade CD19+ malignancy
* No known contraindications to myeloablative HSCT, leukapheresis, steroids or tocilizumab, smallpox vaccine and any other modified vaccinia Ankara (MVA)-based vaccines
* Patient must be CMV seropositive
* Total serum bilirubin =< 2.0 mg/dL
* Participants with Gilbert syndrome may be included if their total bilirubin is =< 3.0
* Aspartate aminotransferase (AST) < 2.5 x upper limits of normal (ULN)
* Alanine aminotransferase (ALT) < 2.5 x ULN
* Serum creatinine =< 2.5 x ULN or estimated creatinine clearance of >= 40 mL/min per the Cockcroft-Gault formula, and the participant is not on hemodialysis
* Absolute neutrophil count >= 1000/uL (Transfusions and growth factors must not be used to meet this requirement at initial screening)
* Hemoglobin (Hb) >= 8 g/dl (Transfusions and growth factors must not be used to meet this requirement at initial screening)
* Platelet count >= 50,000/uL (>= 30,000/uL if bone marrow plasma cells are => 50 percent of cellularity) (Transfusions and growth factors must not be used to meet this requirement at initial screening)
* Left ventricular ejection fraction >= 45 percent within 8 weeks before enrollment
* Oxygen (O2) saturation > 92% without requiring supplemental oxygen
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test
* If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 months after the last dose of protocol therapy.

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Prior autologous/allogeneic stem cell transplant
* Growth factors within 14 days of enrollment
* Platelet transfusions within 7 days of enrollment
* Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled or topical steroids in standard doses is not exclusionary. Physiologic replacement of steroids (prednisone =< 5 mg /day, or equivalent doses of other corticosteroids) is allowed
* Patients with active autoimmune disease requiring systemic immune suppressive therapy are not allowed
* Participants may not be receiving any other investigational agents or concurrent biological therapy, chemotherapy, or radiation therapy
* Any standard contraindications to myeloablative HSCT per standard of care practices at COH
* Subjects with clinically significant arrhythmia or arrhythmias not stable on medical management within two weeks of screening
* Subjects with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system (CNS), including seizure disorder, any measurable masses of CNS, or any other active CNS disease. Note: Research participants with a history of CNS disease that has been effectively treated to complete remission (< 5 white blood cells [WBC] / mm^3 and no blasts in cerebrospinal fluid [CSF]) will be eligible
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agents or cetuximab
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to screening
* History of other malignancies, except for malignancy surgically resected (or treated with other modalities) with curative intent, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; non-muscle invasive bladder cancer; malignancy treated with curative intent with no known active disease present for >= 3 years.
* Clinically significant uncontrolled illness
* Active infection requiring antibiotics
* Immunodeficiency virus (human immunodeficiency virus [HIV]) positive
* Active viral hepatitis
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures
* Procedures (including compliance issues related to feasibility/logistics). Prospective participants who, in the opinion of the investigator, may not be able to comply with all study
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 15 years
  Will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 from data obtained at each clinical assessment. Will be summarized in terms of type (organ affected or laboratory determination), severity, time of onset, duration, probable association with the study treatment and reversibility or outcome.

SECONDARY OUTCOMES:
Achievement of proposed 10×10^6 cytomegalovirus (CMV)-specific CD19-chimeric antigen receptor (CAR) T cells per product and meeting product release requirements for enrolled participants | Up to 56 days
  Yield of at least 10×10^6 cytomegalovirus (CMV)-specific CD19-chimeric antigen receptor (CAR) T cells per product meeting product release requirements
Short- and long-term CMV-specific CD19-CAR T cell expansion and persistence | Up to 15 years
  Will be assessed longitudinally. Persistence is defined as detection of >= 0.1% of CMV-specific CD19-CAR T cells in CD3+ cells in peripheral blood, 28 days after vaccine administration, by flow cytometry and Woodchuck Hepatitis Virus Posttranscriptional Regulatory Element (WPRE) quantitative polymerase chain reaction (Q-PCR). Expansion is defined as an increase of 2-fold in CMV-specific CD19-CAR T cells after Triplex administration compared with pre-vaccination cell number. Response to Triplex will be assessed based on numbers of EGFR+, pp65-specific IFNgamma+ and CD137+T cells.
Clinically significant CMV reactivation | Up to 15 years
  Clinically significant defined as > 1250 IU/ml or 500 GC/mL) CMV reactivation requiring management treatment after CAR T cell infusion as assessed by PCR.
Progression-free survival (PFS) | From the start of treatment to the date of death, disease relapse, or last follow-up whichever occurs first, assessed up to 15 years
  Participants are considered a failure for this endpoint if they die (regardless of cause) or experience disease relapse.
Overall survival (OS) | From start of protocol therapy to death, or last follow-up, whichever comes first, assessed up to 15 years
  Participants are considered a failure for this endpoint if they die, regardless of cause. Will be estimated using the product-limit method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Herrera, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States